CLINICAL TRIAL: NCT05233982
Title: MITO 35a: A Multicenter, Prospective, Single Arm Trial of Olaparib Maintenance Therapy in Newly Diagnosed BRCA Wildtype Advanced Ovarian, Fallopian Tube and Primitive Peritoneal Cancer
Brief Title: MITO 35a: Olaparib Maintenance Therapy in Newly Diagnosed BRCA Wild-type Advanced Ovarian, Fallopian Tube and Primitive Peritoneal Cancer
Acronym: MITO 35a
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2021-000244-21
Record Dates: First submitted 2022-01-18; First posted 2022-02-10 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer
Keywords: olaparib; ovarian cancer; BRCA wilde-type
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OLAPARIB (Experimental)
  Interventions: Drug: Olaparib Oral Product

INTERVENTIONS:
Drug: Olaparib Oral Product — Olaparib Maintenace Treatment after first line platium based chemotherapy in BRCA wilde-type ovarian cancer patients

SUMMARY:
This trial is a multicenter, prospective, phase II single arm, open-label trial in which patients with newly diagnosed advanced epithelial ovarian, primitive peritoneal, and fallopian tube cancer BRCA wild type, in partial or complete response to first line platinum-based chemotherapy, receive Olaparib maintenance therapy (300 mg, tablets formulation twice daily).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained prior to initiation of any study-specific procedures.
2. Female aged≥18 years old on day of signing informed consent.
3. Patients with histologically diagnosed advanced stage III-IV according International Federation of Gynaecology and Obstetrics (FIGO), high grade serous or endometrioid, epithelial ovarian cancer (including primary peritoneal or fallopian tube cancer).
4. Patients with a complete or partial response to first line platinum-based treatment not including Bevacizumab.
5. Documented absence of somatic and germline mutations of BRCA 1 /2.
6. Patients must have a life expectancy ≥ 16 weeks.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1, (See Appendix A).
8. Availability of sufficient formalin-fixed paraffin-embedded (FFPE) tumor tissue from the primary surgery (chemotherapy - naïve patients) for translational analysis. A quality control analysis of samples will be performed before patient's enrollment.
9. Patients must be enrolled within 8 weeks of the first day of the last dose of chemotherapy.
10. Patients must be able to take oral medications.
11. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on Day 1 Cycle 1.

    Postmenopausal is defined as:
    * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments;
    * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50;
    * radiation-induced oophorectomy with last menses >1 year ago;
    * chemotherapy-induced menopause with >1 year interval since last menses;
    * surgical sterilisation (bilateral oophorectomy or hysterectomy).
12. Women Women of childbearing potential and their partners, who are sexually active, must agree to the use of one highly effective forms of contraception and their partners must use a male condom (as described in Appendix D). This should be started from the signing of the informed consent and continue throughout the period of taking study treatment and for at least 1 month after last dose of study drug
13. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

    Haemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days; Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; Platelet count ≥ 100 x 109/L; Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN); Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN

    Patients must have creatinine clearance estimated of ≥51 mL/min using the Cockcroft-Gault equation or based on a 24-hour urine test:
    * Estimated creatinine clearance = (140-age [years]) x weight (kg) (x F) a
    * serum creatinine (mg/dL) x 72 a where F=0.85 for females
14. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Patients have received Bevacizumab in concomitance with first line platinum-based therapy.
2. Clear cell, mucinous and mixed mullerian tumors/carcinosarcoma, non-epithelial tumors or ovarian tumors with low malignant potential (ie. borderline tumors) are not allowed.
3. Received chemotherapy within 14 days to first dose to study drug and / or persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) version 5.0 grade 2) caused by previous cancer therapy, excluding alopecia, peripheral neuropathy and related effects of prior chemotherapy that are unlikely to be exacerbated by treatment with study drug.
4. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
5. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable).
6. Breast feeding women.
7. Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
8. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection [Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, New York Heart Association (NYHA) grade II or greater congestive heart failure, uncontrolled hypertension, severe peripheral vascular disease, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric illness ]
9. Patients with active second malignancy.
10. Other malignancy unless curatively treated with no evidence of disease for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma.
11. Any prior treatment for ovarian cancer, other than first line platinum-based therapy, including any maintenance treatment between completion of the platinum regimen and initiation of study drug in this study.
12. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
13. Concurrent treatment with other investigational agents.
14. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
15. Any positive test result for hepatitis B virus or hepatitis C virus indicating presence of virus, eg. Hepatitis B surface antigen (HBsAg, Australia antigen) positive, or Hepatitis C antibody (anti-HCV) positive (except if HCV-RNA negative).
16. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
17. Patients with symptomatic uncontrolled brain metastases. A TC/RMN scan of brain is required at baseline. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment.
18. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
19. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation < 470 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
20. Evidence of any other medical conditions, physical examination or laboratory findings that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment related complications;
21. Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
22. Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
23. Patients with a known hypersensitivity to olaparib or any of the excipients of the product;
24. Presence of any other condition that may increase the risk associated with study participation or may interfere with the interpretation of study results, and in the opinion of the investigator, would make the

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS). | From date of enrollment until the date of first documentated progression or date of death from any cause, whichever came first, assessed up to 60 months
  PFS as defined by the Investigator using RECIST 1.1 as the time frame from enrollment to progression or death for any cause.

SECONDARY OUTCOMES:
Progression-free survival 2 (PFS2) | From date of enrollment until the date of second documentated progression or date of death from any cause, whichever came first, assessed up to 60 months
  PFS2 as defined by the Investigator using RECIST 1.1, as the time frame from enrollment to the second progression or death for any cause after subsequent treatment.
Overall Survival | 5 years
  OS is defined as the time elapsed from randomization to death due to any cause
Number of participants with treatment-related side effects graded according to Common Criteria for Adverse Events (CTCAE) version 5.0 | At baseline,at end of each cycle (each cycle is 28 days) until progression disease or treatment discontinuation (up to 24 months)]
  Number of participants with treatment-related side effects graded according to Common Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - ONCOLOGIA MEDICA A.O. S. Giuseppe Moscati, Avellino
  - U.O.C. Oncologia Medica - Ospedale Senatore Antonio Perrino, Brindisi
  - IRCCS Istituto Nazionale Tumori di Napoli, Naples
  - Oncologia Medica 2 - Istituto Nazionale Tumori "Regina Elena", Roma
  - ONCOLOGIA MEDICA 1 Istituto Nazionale Tumori Regina Elena - IRCCS - IFO, Rome

REFERENCES:
- See also: Sponsor web-site for study conduction — https://usc.istitutotumori.na.it